CLINICAL TRIAL: NCT01190709
Title: Study of Surgical Methods for Treatment of Tibial Fractures
Brief Title: Study of Tibial Shaft Fracture Fixation: Intramedullary Nailing Comparing With Dynamic Compression Plate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-6
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2008-10

CONDITIONS: Tibial Shaft Fracture
Keywords: Close Fracture; Tibia; Unreamed Intramedullary Nailing; Dynamic Compression Plate
MeSH Terms: conditions — Fractures, Closed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- unreamed Intramedullary Nailing (Other): tibial fracture fixed with unreamed Intramedullary Nailing
  Interventions: Procedure: Unreamed intramedullary nailing
- Dynamic Compression Plate (Other): tibial fracture fixed with Dynamic Compression Plate
  Interventions: Procedure: Dynamic Compression Plate

INTERVENTIONS:
Procedure: Dynamic Compression Plate — we made a longitudinal incision 1 cm lateral to the tibial crest, expose the fracture, and retract the muscles laterally. After determining the length of plate, we used bending instruments to contour the plate to the anatomy then threaded plate holders used to position the plate on the bone. After that we placed the drill guide at the edge of the dynamic compression unit (DCU) portion of the plate hole without applying pressure and tightening of the cortex screws results in dynamic compression. We verified the screw position with a guide wire before insertion and then inserted the locking screw.
  Other Names: DCP
  Arms: Dynamic Compression Plate
Procedure: Unreamed intramedullary nailing — we inserted the nail, without reaming, across the fracture site, with particular attention being paid to the prevention of over distraction and the achievement of cortical contact of the fracture ends. An upper diameter limit of 10 mm and a nail measuring at least 2 mm less than the diameter measured at the isthmus of the tibia on anteroposterior and lateral radiographs were stipulated.
  Other Names: DCP
  Arms: unreamed Intramedullary Nailing

SUMMARY:
The purpose of this study is to determine which surgical approach is better for treatment of tibial shaft fracture

DETAILED DESCRIPTION:
Tibial fracture is more common fracture. We aimed to compare unreamed intramedullary nailing (UTN) and dynamic compression plate (DCP) with regard to fracture healing and complications in patients with closed tibial shaft fractures.

ELIGIBILITY:
Inclusion Criteria:

* patient with tibial shaft fracture

Exclusion Criteria:

* nothing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
time of fracture healing | at 16 months post-operatively
  identification of time of fracture healing in patients who underwent plate or nail methods

SECONDARY OUTCOMES:
malunion | at 16 months post-operatively
  identification of rate of malunion in two surgical groups
nonunion | at 16 months post-operatively
  identification of rate of nonunion in two surgical groups
infection | at 16 months post-operatively
  identification of rate of infection in two surgical groups

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran